CLINICAL TRIAL: NCT03330210
Title: National Longitudinal Registry for Mid-Term Clinical Outcome And Procedure Efficacy Evaluation In Using A Novel Preprocedural Planning Method For Left Atrial Appendage Occlusion Guided By 3D Printing
Brief Title: Left Atrial Appendage Occlusion Guided by 3D Printing
Acronym: LAA-PrintRegis
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hôpital Privé Les Franciscaines (Other); Henri Mondor University Hospital (Other); Rangueil Hospital (Other); Clinique Pasteur Toulouse (Other); University Hospital, Bordeaux (Other); Clinique du Millenaire (Other); Clinique Saint Pierre - Perpignan (Unknown); Hôpital Dupuytren (Other); Hospital St. Joseph, Marseille, France (Other); European Georges Pompidou Hospital (Other); University Hospital, Grenoble (Other); University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0230
Record Dates: First submitted 2017-10-11; First posted 2017-11-06 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: LAAC; 3D printing; Procedure success; Procedure-related complications
MeSH Terms: conditions — Atrial Fibrillation | interventions — Printing, Three-Dimensional

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: 3D printing — Manufacturing and use of a model printed in 3D

SUMMARY:
Left atrial appendage closure (LAAC) was approved by the ESC guidelines as a stroke prevention alternative to warfarin for patients with nonvalvular atrial fibrillation in patients at high risk of bleeding (IIbB).

Although the overall LAAC benefice, in term of prevention of stroke or embolisme and decresing the anticoagulant-related risk of bleeding is already demonstrated, however the procedure success and safety, critically depends on understanding LAA anatomy and adequate pre-procedure planning.

3D-printed patient-specific adaptive and flexible LA models have demonstrated in a previous study an improving in LAAO device sizing, a better pre-procedural planning of the optimal trans-septal puncture site, by incorporating all anatomical variations and an improuving patient outcomes by reducing procedure time and number of prostheses employed per patient.

This technique is now used in several surgical centers in France and large prospective evaluation of the practice is necessary.

DETAILED DESCRIPTION:
The 3D printing has modified the LAAC practices with a preoperative time allowing an optimal preparation of the prosthesis. This technique is now used in several surgical centers and prospective evaluation of the practice is necessary.

The objective of our research is to demonstrate the reduction of the operating time and number of prosthesis used per procedure when prior LAAC simulation testing and sizing is made on a 3D printed model.

It is therefore a longitudinal research to monitor professional practices for the evaluation of a new preoperative approach.

Procedures guided by 3Dprinted models will be compared (intention to treat population) in term of procedural parameters (procedure time, success rate, number of prosthesis per procedure) and procedural complication with prior Watchman study: post-FDA Approval US experience and national registries data. A second analysis (per protocol population) will be performed to compare patients with an informative utilization guided by 3D printed to those of the post-FDA Approval US experience and national registries.

ELIGIBILITY:
Inclusion Criteria:

* non valvular AF
* adressed for LAAC procedure

Exclusion Criteria:

* opposition from patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in atrial fibrillation addressed for percutaneous left atrial appendage closure intervention
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
operating time | During 1 day
  mesure of operating time to Day 0 (J0)
number of protheses | During 1 day
  decrease number of prothèses to Day 0 (J0)
Implantation success rate | During 1 day
  increase implantation success rate at Day 0 (J0)

SECONDARY OUTCOMES:
number of periprosthetic leak | During 1 day
  decrease number of periprosthetic leak at Day 0 (J0)
anasthesia time | During 1 day
  decrease of anasthesia time at Day 0 (J0)
time of scopy | During 1 day
  decrease time of scopy at Day 0 (J0)
irradiation dose | 1 day
  decrease of irradiation dose (mGy.cm2) at Day 0 (J0)
Days of Hospitalisation | During 1 day
  discharge and decrease of hospitalisation days
number of recapture | During 1 day
  decrease number of recapture at Day 0 (J0)
number of off-axis prostheses | During 1 day
  decrease number of off-axis prosthèses at Day 0 (J0)
number of embolized prostheses | During 1 day
  decrease number of embolized prosthèses at Day 0 (J0)
Effective complete occlusion of the auricle | 3 months
  increase rate of Effective complete occlusion of the auricle
Effective complete occlusion of the auricle | 6 months
  increase rate of Effective complete occlusion of the auricle
prosthesis trombosis | 12 months
  rate of prosthesis trombosis
procedural complications | during procedure and within 30 days
  analysis of complications (Stroke, transient ischaemic attack, peripheral embolism, Pericardial effusion and tamponade Bleeding, Life threatening, major and minor, Acces related complications, Renal or hepatic acute failure)
complication | 6 and 12 months
  analysis of complications (Stroke, transient ischaemic attack, peripheral embolism, Pericardial effusion and tamponade Bleeding, Life threatening, major and minor, Acces related complications, Renal or hepatic acute failure) at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vlad CIOBOTARU, Study Chair — Hôpital Privé Les Franciscaines
Locations (1):
- Hôpital Privé les Franciscaines, Nîmes, France